CLINICAL TRIAL: NCT01716364
Title: A Phase I Study Investigating Safety Immunological Effects of Peripheral Blood T Lymphocytes Transduced With Anti LewisY Chimeric Receptor Gene in LewisY Positive Myeloma, Acute Myeloid Leukemia or High Risk Myelodysplastic Syndrome
Brief Title: Safety Study of Anti LewisY Chimeric Antigen Receptor in Myeloma, Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LeYPh1
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-10

CONDITIONS: Multiple Myeloma; Acute Myeloid Leukaemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anti-LeY- scFv-CD28-ζ vector. (Experimental): Anti-LeY- scFv-CD28-ζ vector, a non-pathogenic, replication-incompetent retroviral vector specifically designed for this study and produced by EUFETS under GMP-conditions.
  Interventions: Biological: Anti-LeY- scFv-CD28-ζ vector,.

INTERVENTIONS:
Biological: Anti-LeY- scFv-CD28-ζ vector,.

SUMMARY:
Patients with some forms of acute myeloid leukemia (AML) and multiple myeloma (MM) are not cured with conventional therapy and new approaches are needed. For the last 15 years we have investigated the potential of using a patient's own T cells (a type of white blood cell [WBC]) to eradicate the tumor. We have demonstrated the feasibility of this approach in cell culture and animal models of AML and MM. Over the last 5 years we have been preparing to treat patients as part of a Phase I (first in human) clinical trial.

The trial treatment involves collecting the patient's own WBCs from the blood by a standard well established and safe process called apheresis. The cells are then cultured in a specialized laboratory (under Good Manufacturing Practice conditions, similar to standards under which pharmaceuticals are produced) over 12 days to convert the cells to specialized tumor-attacking T cells. Early in that culture process the cells are exposed to a virus (that is modified so that it cannot infect or replicate outside the special culture conditions) that contains a special gene. Via the virus, this gene inserts into the patient's T cells in culture and gets incorporated into the T cell's genetic machinery. As the T cells replicate, the new gene produces a protein receptor that becomes part of the patient's T cells. This protein receptor on the T cells has the capacity to specifically recognize and bind to a protein on the leukemia or myeloma cells called the "Lewis Y" antigen.

After the modified T cells are infused into the patient, they home into the bone marrow (this tracking is monitored by special radiological techniques) where the new protein receptor on the T cell surface can recognize and bind to the cancer cells (which express Lewis Y). Once bound onto the cancer cells, the T cells get activated and subsequently replicate and kill the cancer cells. The novelty of this approach is that the T-cells will only kill cells that have the Lewis Y on their surface - the cancer cells. Moreover, because there are few normal cells in a person's body that carry Lewis Y, this treatment is likely to only have minor side effects.

This gene therapy trial is unique and although the primary purpose is to test the safety of this approach, patients will be monitored closely for anti-tumor responses. As the trial progresses, the dose of T cells infused will increase, in the hope that this will result in a better and stronger immune response to the leukemia or myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Applicable to all Patients
* Patient is able to undergo apheresis of peripheral blood mononuclear cells (PBMC) within eight weeks following registration.
* White cell count (WCC) <30/nL as higher WCC could interfere with the apheresis of PBMC.
* Patient has an ECOG performance status of 0 - 1.
* Patient is deemed capable of undergoing the planned study procedures
* Patient has adequate organ function:

  * bilirubin <1.5x upper limit of normal (ULN), AST/ALT ≤2.5 x ULN except in patients with Gilbert's syndrome
  * Serum Creatinine < 1.5 ×ULN or creatinine clearance > 50ml/min
  * Amylase, lipase ≤1.5xULN
* Lymphocyte count of ≥0.5x109/L
* > 18 years of age.
* Patient has provided written informed consent.
* No chemotherapy or treatment with G-CSF within 4 weeks prior to the planned apheresis.
* Applicable to patients with multiple myeloma
* Patient has histologically or cytologically confirmed diagnosis of multiple myeloma plus one or more of the criteria set out below must apply:
* Presence of the following features that are known to be associated with an adverse prognosis with conventional chemotherapy, high-dose chemotherapy and autologous stem cell transplant (AUSCT):

Chromosomal abnormalities:

* 13q deletion
* 17p deletion as p53-deletion by IHC on the bm trephine
* Translocation (4:14)
* Translocation (14:16)

Clinical features:

* Progressive disease within 12 months after previous AUSCT
* Plasmablastic morphology
* Plasma cell leukaemia

  * Patient planned for high-dose melphalan chemotherapy with AUSCT having had at least two prior treatment regimens (which can include prior high-dose chemotherapy and AUSCT and must include at least one of thalidomide, lenalidomide or bortezomib).
  * Patient has previously proven LewisY expression on the plasma cells prior to study entry in an analysis as defined in study criteria
  * Patient is planned to receive high dose melphalan and autograft (after apheresis of PBMC)
  * Additional inclusion Criteria applied to patients with acute myeloid leukaemia (AML)/high-risk myelodysplastic syndrome (MDS)

All of the following must apply:

* Patient must either have newly diagnosed AML/high-risk MDS with a poor prognosis or relapsed/refractory AML/high-risk MDS
* Patient has previously proven LewisY expression on the myeloblasts prior to study entry in an analysis as defined in study criteria
* Patient is planned to receive fludarabine containing regime (FCR) chemotherapy (after apheresis of PBMC) which is planned to be the last cycle of FCR chemotherapy, no further FCR chemotherapy should be planned within 3 months after this cycle of FCR

Definition of poor prognosis in AML/high-risk MDS

A patient with AML has a poor prognosis if any of the following is satisfied:

* Age > 65 years
* Age 56 - 65 years with any of the following single cytogenetic abnormalities: -7, -5, trisomy 8, abnormal 3q, t(6;9), t(9;22) or t(9;11), normal karyotype with FLT3-ITD
* Age 56 - 65 years with a complex aberrant karyotype defined as >4 cytogenetic abnormalities
* Any age with relapsed or refractory disease

Exclusion Criteria

None of the following should apply:

* Patient has had immunotherapy including corticosteroids (except Prednisolone <10mg or equivalent) within the last 4 weeks or is planned to receive such therapy prior to apheresis of PBMC.
* Patient has been given chemotherapy and/or G-CSF in the last 4 weeks.
* Patient has been planned to receive chemotherapy and/or growth factors of any type before planned apheresis of PBMC
* Patient has been given experimental therapy within the last 4 weeks or is planned to receive experimental therapy prior to apheresis of PBMC
* Patient has known clinically significant autoimmune disease with positive serology for RHF (>20kU/L) or ANA (titre >1:40)
* Patient has a history of idiopathic pancreatitis Patient has known, biopsy proven autoimmune inflammatory disease of the gastrointestinal tract
* Women of child bearing potential (WOCBP) who are unwilling or unable to use an effective method of contraception to avoid pregnancy for the entire study period and for at least 3 months after completion of study treatment.
* Women who are pregnant or breastfeeding.
* Men who are unwilling or unable to use an acceptable method of contraception for the entire study period and for at least 3 months after completion of study treatment if their sexual partners are WOCBP.
* Patient has known central nervous system (CNS) disease.
* Patient has a serious uncontrolled medical disorder which would impair the ability to receive protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events. | Up to 3 years

SECONDARY OUTCOMES:
Percentage of infused labelled cells localizing in bone marrow | Up to 3 years
Percentage of infused labelled cells localizing in soft tissue or plasmacytoma. | Up to 3 years
Presence or absence of anti-LeY positive T-cells in peripheral blood and bone marrow. | Up to 3 years
Percentage of anti LeY positive T-cells in peripheral blood and bone marrow. | Up to 3 years
Serum IFN-γ and IL-2 levels. | Up to 3 years
Presence or absence of autoimmune disease. | Up to 3 years
Overall response. | Up to 3 years
Time to progression | Up to 3 years
Time to treatment failure | Up to 3 years
Duration of response | Up to 3 years
Overall survival | Up to 3 years
Location of labelled re-infused T-cells | Up to 1 month
LewisY expression assessed with Flow Cytometry in Peripheral Blood and Bone Marrow. | Up to 3 years
LewisY expression assessed with Flow Cytometry in Peripheral Blood and Bone | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Miles Prince, MD, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia